CLINICAL TRIAL: NCT06571305
Title: FAMILY Sleep Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Community Foundation for Brevard (Unknown)
Responsible Party: Principal Investigator, Youngmee Kim, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20231290; NCI-2024-06704 (Registry Identifier: NCI Clinical Trials Reporting Program (NCI CTRP))
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 2 BBTI Intervention Group (Experimental): Participants (patient-sleep-partner caregiver dyads) in this group will receive the Brief Behavioral Treatment for Insomnia (BBTI). Total participation is up to 4 weeks.
  Interventions: Behavioral: Brief Behavioral Treatment for Insomnia (BBTI)
- Phase 2 MSOS Intervention Group (Experimental): Participants (patient-sleep-partner caregiver dyads) in this group will receive the My Sleep Our Sleep (MSOS) intervention. Total participation is up to 4 weeks.
  Interventions: Behavioral: My Sleep Our Sleep (MSOS)

INTERVENTIONS:
Behavioral: Brief Behavioral Treatment for Insomnia (BBTI) — BBTI is brief patient-focused intervention for patient-sleep-partner caregiver dyads, aimed at altering participants' sleep behaviors to improve sleep. BBTI utilizes behavioral education in sleep restriction and stimulus control. For sleep restriction, participants will be instructed to limit the time spent in bed, which serves to increase sleep efficiency. For stimulus control, participants will be instructed to go to bed only when feeling sleepy and reserve the bed for sleep and intimacy.
  BBTI will be delivered over four weeks, in weekly one-hour sessions, one session per week.
  Arms: Phase 2 BBTI Intervention Group
Behavioral: My Sleep Our Sleep (MSOS) — MSOS is a sleep intervention developed by the investigator aimed at improving sleep health for patient-sleep-partner caregiver dyads using behavioral education in sleep behaviors, sleep cognition and sleep in relationship.
  MSOS will be delivered over four weeks, in weekly one-hour sessions, one session per week.
  Arms: Phase 2 MSOS Intervention Group

SUMMARY:
The purpose of this study is to learn about sleep behaviors and test different ways to help patients with cancer and partners. Participants (patient-sleep-partner caregivers dyads as a unit) participate in the study together.

ELIGIBILITY:
Inclusion Criteria:

* The eligibility criteria for patients are

  * newly diagnosed with stage I to IV of a solid tumor
  * diagnosis in the past seven years at the time of enrollment
  * having a consistent sleep partner.
* The eligibility criterion for caregivers is

  * a sleep partner of the patient.
* Additional eligibility criteria for both patients and caregivers are

  * Pittsburgh Sleep Quality Index (PSQI) ≥ 5,
  * willing to change sub-optimal sleep habits,
  * 18 years or older,
  * able to speak/listen English at the 8th grade level for intervention sessions,
  * able to read English or Spanish at the 8th grade for self-reported questionnaires, reside in Brevard County, Florida (FL),
  * only for participants of Aim 2, > 4 weeks after surgery, if any, prior to enrollment, and no surgery planned in the next 5 weeks during the study period because surgery affects sleep.

Exclusion Criteria:

* Exclusion criteria for both patients and caregivers are:

  * having had a diagnosis of major depressive disorder, psychosis, or bipolar disorder that is not currently treated;
  * active suicidality, or substance or alcohol dependency in the past year;
  * currently have narcolepsy, restless leg syndrome, or untreated sleep apnea that is screened using the Sleep Health Screen;
  * both patients and caregivers have an extreme chronotype, or do shift work to have no overlap in sleep schedule between them; and
  * plan trans-meridian travel during the period of data collection blocks; and
  * having hearing or visual impairment, dementia, or cognitive dysfunction.
* Adults unable to consent, individuals who are not yet adults, pregnant women, or prisoners will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants adapting to BBTI | Up to 4 weeks
  The proportion of participants (patient--sleep-partner caregiver dyads) who adapt to Brief Behavioral Treatment for Insomnia (BBTI).
Change in Sleep Disturbance Symptoms Measured by Pittsburgh Sleep Quality Index (PSQI) | Baseline, Up to 4 weeks
  The proportion of participants (patient-sleep-partner caregiver dyads) experiencing a change in sleep disturbance symptoms will be compared and reported for both intervention groups, BBTI and MSOS, as measured by scores on the Pittsburgh Sleep Quality Index (PSQI) health-related quality of life HRQOL) questionnaire. The PSQI is a self-reported, 19-item questionnaire which assesses sleep quality and disturbances at baseline and over a four week period. Questions generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score. The PSQI global score has a possible range of 0-21 points. A total score of 5 or above indicates overall poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Youngmee Kim, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No